CLINICAL TRIAL: NCT05430724
Title: The Effects of Nicardipine and Esmolol Applied for Controlled Hypotension in Rhinoplasty Procedures on Hemodynamics and Regional Renal Oxygenation
Brief Title: The Effects of Nicardipine and Esmolol Applied for Controlled Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Assoc. Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Controlled hypotension esmolol
Record Dates: First submitted 2022-05-12; First posted 2022-06-24 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Hypotension; Surgery-Complications; Oxygen Deficiency
Keywords: Controlled hypotension; rhinoplasty; esmolol; nicardipine; regional renal oxygenation
MeSH Terms: conditions — Hypotension; Hypoxia

STUDY DESIGN:
Intervention Model Description: The patients included in the study will be divided into 2 groups according to the closed envelope system. Patients given esmolol infusion will be named Group E (n:40), patients given nicardipine infusion will be named Group N (n:40).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup E (Active Comparator): Patients given esmolol infusion
  Interventions: Procedure: Controlled hypotention
- Grup N (Active Comparator): Patients given nicardipine infusion
  Interventions: Procedure: Controlled hypotention

INTERVENTIONS:
Procedure: Controlled hypotention — The procedure to be applied to the cases to be included in the study:
  Patients randomized by the sealed envelope method will be divided into 2 groups (40 patients in each group).
  The sealed envelopes that determine which group the patient will belong to will be randomly selected by the patient.
  Standard general anesthesia will be applied to all patients. Before starting the surgical procedure; Group N (Nicardipine infusion) will be administered at a dose of 5-15mg/h, and Group E (Esmolol infusion) at a dose of 50-300mcg/kg/min.
  2) General anesthesia will be applied to all groups. Patients will be administered controlled hypotension (mean arterial pressure 50-60 mmHg).

SUMMARY:
In this study, the effects of nicardipine and esmolol applied for controlled hypotension in rhinoplasty on hemodynamics and regional renal oxygenation will be investigated.

DETAILED DESCRIPTION:
The procedure to be applied to the cases to be included in the study:

Patients randomized by the sealed envelope method will be divided into 2 groups (40 patients in each group).

The sealed envelopes that determine which group the patient will belong to will be randomly selected by the patient.

Standard general anesthesia will be applied to all patients. Before starting the surgical procedure; Group N (Nicardipine infusion) will be administered at a dose of 5-15mg/h, and Group E (Esmolol infusion) at a dose of 50-300mcg/kg/min.

2) General anesthesia will be applied to all groups. Patients will be administered controlled hypotension (mean arterial pressure 50-60 mmHg).

After the patients are taken to the operating table, standard electrocardiography (ECG), peripheral oxygen saturation (SpO2), heart rate (HR), blood pressure monitoring, and regional renal oxygenation will be provided with Near-infrared reflectance spectroscopy (NIRS) monitoring. .

Systolic arterial pressure (SAB), diastolic arterial pressure (DAP), mean arterial pressure (MAP), HR, SpO2, and NIRS values will be recorded.

3) Demographic data of the patients [age, weight, height, body mass index (BMI), smoking], duration of operation, need for intraoperative muscle relaxants and/or opioids, surgical satisfaction and intraoperative blood loss will be recorded.

4) General anesthesia procedure: After monitoring as standard, vascular access will be opened with 2 pieces of 18 gauge cannula. After adequate preoxygenation, induction will be achieved with 2mg/kg propofol, 2/µg fentanyl and 0.6mg rocuronium. In the maintenance of anesthesia, 40% O2, 60% medical air and 1 MAC value Desflurane inhaler will be used as anesthetic agent. Anesthesia puberty will be followed by BIS monitoring and BIS value will be kept between 40-60 in all patients.

For regional renal oxygenation, NIRS probes will be placed in both kidneys (at the level of the posterior axillary line, between the lumbar 6-7 range. After the initial value is recorded, recordings will be taken every 5 minutes throughout the operation. A 20% change in values will be considered significant.

At the end of the operation, after standard decurarization, extubation will be performed when appropriate conditions are met. After the recovery, the Mini Mental Test will be filled in the patient.

A surgical satisfaction questionnaire will be filled after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-60 years of age,
* ASA I-II,
* undergoing elective rhinoplasty surgery,
* it was decided to apply controlled hypotension,
* BMI (body mass index) between 18-25 kg/m2,
* informed about the subject and
* patients with written consent

Exclusion Criteria:

* ASA III-IV patients,
* hypertension disease,
* using anticoagulant medication,
* pregnancy,
* kidney failure,
* bleeding diathesis,
* active infection,
* allergy to drugs to be used,
* BMI≥30,
* refusing to participate in the study,
* hypothermic,
* patients taking antibiotics, anticonvulsants, antiarrhythmics, cholinesterase inhibitors

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Level of hypotension | 1 year
  Measuring mean blood pressures
Monitoring of renal oxygen saturation | 1 year
  Measurement of regional renal oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yuzkat, Principal Investigator — Van Yuzuncu Yil University, Faculty of Medicine, Tusba, Van, Turkey
Locations (1):
- Van yuzuncu Yıl University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan wil be share other researchers
Supporting Information: Study Protocol, SAP
Time Frame: One year
Access Criteria: the access can be provided via the e-mail addresses below nyuzkat@gmail.com

REFERENCES:
- [Background] Lin S, McKenna SJ, Yao CF, Chen YR, Chen C. Effects of Hypotensive Anesthesia on Reducing Intraoperative Blood Loss, Duration of Operation, and Quality of Surgical Field During Orthognathic Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Oral Maxillofac Surg. 2017 Jan;75(1):73-86. doi: 10.1016/j.joms.2016.07.012. Epub 2016 Jul 25. PMID 27542543
- [Result] Pilli G, Guzeldemir ME, Bayhan N. Esmolol for hypotensive anesthesia in middle ear surgery. Acta Anaesthesiol Belg. 1996;47(2):85-91. PMID 8869676
- [Result] Steppan J, Hogue CW Jr. Cerebral and tissue oximetry. Best Pract Res Clin Anaesthesiol. 2014 Dec;28(4):429-39. doi: 10.1016/j.bpa.2014.09.002. Epub 2014 Sep 28. PMID 25480772